CLINICAL TRIAL: NCT05488548
Title: A Phase 1 Study of EP31670, a Dual BET and CBP/p300 Inhibitor in Patients With Targeted Advanced Solid Tumors and Hematological Malignancies
Brief Title: Dual BET and CBP/p300 Inhibitor in Patients With Targeted Advanced Solid Tumors and Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Epigenetix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP31670-01
Record Dates: First submitted 2022-07-27; First posted 2022-08-04 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-09

CONDITIONS: Castrate Resistant Prostate Cancer; NUT Carcinoma; Chronic Myelomonocytic Leukemia; Myelofibrosis
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Primary Myelofibrosis | interventions — NEO2734

STUDY DESIGN:
Intervention Model Description: Dose escalation/de-escalation will follow rules by employing the Bayesian optimal interval (BOIN) method for Part 1 and Part 2 and traditional 3+ 3 by modified Fibonacci sequence for Part 3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Patients will be assigned escalated dose according to BOIN design. The starting dose is 5 mg orally once a day for 7 consecutive days followed by 14 days of rest.
  Interventions: Drug: EP31670
- Part 2 (Experimental): Patients will be assigned escalated dose according to BOIN design. The starting dose is 20 mg orally once a day for 14 consecutive days followed by 14 days of rest.
  Interventions: Drug: EP31670
- Part 3 (Experimental): Patients will be assigned escalated dose according to BOIN design. The starting dose is 10 mg orally once a day for 14 consecutive days in combination with ruxolitinib or momelotinib followed by 14 days of rest according to the traditional 3 + 3 design by the modified Fibonacci sequence
  Interventions: Drug: EP31670

INTERVENTIONS:
Drug: EP31670 — EP31670 (also known as NEO2734) is a first-in-class dual BET and CBP/p300 inhibitor.
  Other Names: NEO2734

SUMMARY:
A Phase 1, first-in-human study of EP31670, a dual BET and CBP/p300 inhibitor in patients with targeted advanced solid tumors and Hematological Malignancies

DETAILED DESCRIPTION:
EP31670 (also known as NEO2734) is a first-in-class dual BET and CBP/p300 inhibitor which has demonstrated antitumor activity in in vitro and in vivo models of human cancer. This Phase I open-label, multi-center, dose-escalation study will assess the safety and determine the maximum tolerated dose of EP31670 administered orally in patients with castration-resistant prostate cancer, NUT midline carcinoma and other targeted advanced solid tumors as well as chronic myelomonocytic leukemia (CMML), myelofibrosis (MF) and other targeted hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Relapse or refractory castration-resistant prostate cancer (CRPC) following at least one anti-androgen regimen and a docetaxel-containing regimen OR
* metastatic or unresectable NUT midline carcinoma for which standard curative or palliative measures do not exist; OR

Part 2

* relapsed or refractory CMML following at least 4 cycles of hypomethylating agent-containing regimen or hydroxyurea unless demonstration of progression or intolerance;
* advanced MF (intermediate or high-risk) following at least one JAK inhibitor-containing regimen or unsuitable candidates for JAK inhibitor treatments.

Part 3: advanced MF (intermediate or high-risk) with ≤10% blasts in peripheral blood who have not achieved an adequate response or have lost the response to a JAK inhibitor-containing regimen after being on treatment for at least 3 months.

Patients who have other types of relapsed or refractory solid tumors (Part 1) or hematological malignancies (Part 2) with pathological and/or biological features suggesting a potential benefit from dual BET and CBP/p300 inhibition may be enrolled after discussion with and approval from medical monitor and sponsor.

Eastern Cooperative Oncology Group (ECOG) performance status 0-1 Life expectancy ≥ 3 months Evaluable disease

Adequate bone marrow function:

* Hemoglobin ≥ 9.0 g/dL (Part 1)
* Absolute neutrophil count (ANC) ≥ 1,500/dL (Part 1)
* Platelet count ≥100,000/μL (Part 1) or ≥75,000/μL (Part 3)

Adequate renal function: Creatinine clearance (CLcr) ≥ 60 mL/min

Adequate liver function: total bilirubin ≤ 1.5 x ULN; alanine aminotransferase (ALT) or aspartate Aminotransferase (AST) ≤ 2.5 x ULN or ≤ 5 x ULN in patients with liver metastases

Internal normalized ratio for prothrombin time (INR) ≤ 1.2 in patients not receiving chronic anticoagulation

Four weeks from prior anti-cancer therapy including chemotherapy, immunotherapy, investigational anti-cancer therapy or 5 half-lives from targeted agents, radiation and have recovered from prior treatment toxicities to grade 1 or less.

Four weeks from major surgery.

For fertile men and women, agreement to use effective contraceptive methods duration of study participation and 4 weeks after the last dose of study drug.

Ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* New and progressive central nervous system (CNS) metastasis; patients with treated brain metastases are eligible if follow-up brain imaging at least 4 weeks after CNS-directed therapy shows no evidence of progression and the patient is neurologically stable
* Corrected QT interval ≥470 msec
* Uncontrolled concurrent illnesses including, but not limited to, ongoing active infection requiring intravenous antibiotics or antifungal agents, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would affect compliance with study requirements; patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of EP31670 are eligible for this trial
* Pregnant or lactating women
* Known history of hepatitis B, hepatitis C requiring antiviral treatment
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within 3 weeks (one cycle) of treatment
  MTD is the highest dose level at which ≤30% of patients experienced DLTs during cycle 1.
Dose Limiting Toxicities (DLT) | Within 3 weeks (one cycle) of treatment
  DLT is any of the following adverse events (AEs) that occur during cycle 1.
Recommended Phase 2 Dose (RP2D) | through study completion, an average of 1 year
  RP2D will be the MTD

CONTACTS AND LOCATIONS:
Overall Officials: Judy Chiao, MD, Study Director — Epigenetix, Inc.
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- [Derived] Eickhoff N, Bergman AM, Zwart W. Homing in on a Moving Target: Androgen Receptor Cistromic Plasticity in Prostate Cancer. Endocrinology. 2022 Oct 11;163(11):bqac153. doi: 10.1210/endocr/bqac153. PMID 36125208